CLINICAL TRIAL: NCT00689572
Title: New Medication Treatment for Stimulant Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nassima Ait-Daoud Tiouririne, Associate Professor, Director of UVA Center for Addiction Research and Education, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13419; 1R01DA021776-01A1 (NIH)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-08

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; cocaine abuse; cocaine; crack
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ondansetron; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ondansetron (Experimental): Ondansetron + Cognitive Behavioral Therapy + Brief Behavioral Enhancement Therapy
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo + Cognitive Behavioral Therapy + Brief Behavioral Enhancement Therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — 4 mg twice a day + Cognitive Behavioral Therapy + Brief Behavioral Enhancement Therapy
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo — twice a day + Cognitive Behavioral Therapy + Brief Behavioral Enhancement Therapy
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of ondansetron compared with placebo in the treatment of cocaine dependence.

DETAILED DESCRIPTION:
We propose to conduct a 9 week randomized, controlled clinical trial to evaluate the efficacy of ondansetron 4 mg twice daily compared with placebo (total N = 100/group × 2 groups = 200 individuals randomized, 400 total subjects will be consented), provided as an adjunct to manual-driven, structured CBT + BBCET in the treatment of cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent.
* Ages 18 years and above and, must weigh at least 40 Kg and no more than 140 Kg.
* Good physical health as determined by a complete physical examination, an EKG within normal limits, and laboratory screening tests within acceptable parameters.
* Current DSM-IV diagnosis of cocaine dependence.
* At least one positive urine drug screen for cocaine at screen or baseline prior to randomization.
* The pregnancy test for females at intake must be negative.
* Literacy in English and ability to read, understand, and complete the ratings scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments.
* Answered an advertisement in the newspaper/radio/television, and expressing a wish to stop using cocaine.
* Willing to participate in behavioral treatments for cocaine dependence.

Exclusion Criteria:

Please contact site for additional information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassima Ait-Daoud Tiouririne, M.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Center for Addiction Research and Education, Charlottesville, Virginia
  - University of Virginia Center for Addiction Research and Education, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blevins D, Seneviratne C, Wang XQ, Johnson BA, Ait-Daoud N. A randomized, double-blind, placebo-controlled trial of ondansetron for the treatment of cocaine use disorder with post hoc pharmacogenetic analysis. Drug Alcohol Depend. 2021 Nov 1;228:109074. doi: 10.1016/j.drugalcdep.2021.109074. Epub 2021 Sep 24. PMID 34600264
- See also: (UVA CARE Website) — https://med.virginia.edu/uva-clear/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ondansetron | Placebo
Started | 53 | 55
Completed | 39 | 34
Not Completed | 14 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron | Placebo | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 55 | 108
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 33 | 33 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 12 | 9 | 21
  American Indian or Alaskan Native | 0 | 0 | 0
  Asian American or Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 45 | 85
  Hispanic | 0 | 0 | 0
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use by Self-report
Description: Participants were assessed up to three times weekly for up to 9 weeks to evaluate cocaine use by self-report
Time Frame: up to 9 weeks
Population: All participants who completed at least one randomly allocated treatment visit were included in the intent-to-treat population.
Measure: Mean (Standard Deviation); unit: Percent of cocaine-free (abstinent)days
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 53 | 55
Percent of cocaine-free (abstinent)days | 67 (0.25) | 67 (0.22)
Statistical Analysis 1: Comparison: Ondansetron vs Placebo; Difference between ondansetron and placebo groups regarding percentage of cocaine-free days (PCFD); Test type: Equivalence — Mixed-effects linear regression model; p = 0.972, Regression, Linear; Mixed-effects linear regression model included random intercept and slope (for temporal trend); Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-5.43 to 5.25]

2. Primary Outcome: Cocaine Use by Urine Benzoylecgonine
Description: Urine samples were collected up to three times weekly for up to 9 weeks to test for the major cocaine metabolite benzoylecgonine
Time Frame: up to 9 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of cocaine-free urines
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 53 | 55
Percent of cocaine-free urines | 16 (0.32) | 26 (0.33)
Statistical Analysis 1: Comparison: Ondansetron vs Placebo; Difference between ondansetron and placebo groups regarding percentage of cocaine free urines (PCFU); Test type: Equivalence — Mixed-effects linear regression model; p = 0.909, Regression, Linear; Mixed-effects linear regression model included random intercept and slope (for temporal trend); Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-7.08 to 7.95]

ADVERSE EVENTS:
Time Frame: up to 9 weeks
Arm/Group | Ondansetron | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/55
Other Adverse Events (participants affected / at risk) | 44/53 | 47/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron (N=53) | Placebo (N=55)
Hospitalization for gallstone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hospialization for stab wound to chest (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansetron (N=53) | Placebo (N=55)
Abdominal Pain (Gastrointestinal disorders) | 19 | 14
Anxiety (Psychiatric disorders) | 7 | 11
Appetite Increase (Gastrointestinal disorders) | 18 | 12
Appetite Decrease (Gastrointestinal disorders) | 18 | 17
Constipation (Gastrointestinal disorders) | 34 | 16
Diarrhea (Gastrointestinal disorders) | 16 | 25
Dizziness (Nervous system disorders) | 5 | 9
Fatigue (Nervous system disorders) | 26 | 13
Headache (Nervous system disorders) | 23 | 24
Insomnia (Nervous system disorders) | 18 | 24
Vomiting (Gastrointestinal disorders) | 13 | 11
Weight Decrease (Metabolism and nutrition disorders) | 3 | 2
Weight Increase (Metabolism and nutrition disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 10
Paresthesia (Nervous system disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Depression (Psychiatric disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 15 | 14
Somnolence (Psychiatric disorders) | 21 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No